CLINICAL TRIAL: NCT05621928
Title: Effectiveness of Vaccination Against COVID-19 in Brazil: Case-Control Study
Status: Active, not recruiting | Type: Observational
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Other Study IDs: 003/2021
Record Dates: First submitted 2022-11-17; First posted 2022-11-18 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — oral and nasopharyngeal secretion, blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- cases with positive RT PCR result for Covid 19: Individuals aged 18 years or older, with a suspected clinical picture of COVID-19 virologically confirmed, that is, with positive RT-PCR for SARS-CoV-2 in a respiratory secretion sample collected in the first 7 days of the onset of symptoms , who did not have a positive RT-PCR result for SARS-CoV-2 in the 90 days preceding enrollment in the study.
- Control: Individuals residing in the vicinity of the case, aged 18 years or older, without a suspected clinical picture of COVID-19 and with RT-PCR negative for SARS-CoV-2 in a respiratory secretion sample collected at the time of inclusion, followed by confirmation of the absence of signs and symptoms suggestive of COVID-19 within the next 7 days.
- immunogenicity analyzes: a convenience sample composed of all cases exposed or not to vaccination and 200 controls, 100 vaccinated and 100 unvaccinated, for analysis of humoral response.
- assessment of cellular immunity: a sample of 100 vaccinated cases and 100 unvaccinated cases followed prospectively, and 100 vaccinated controls 100 unvaccinated controls assessed spot-on at enrollment.
- analysis of potential genetic risk factors for the occurrence of severe forms of COVID-19 (SRAG): a total of 50 cases

SUMMARY:
The main objective of the study is to evaluate the effectiveness of the vaccine against covid-19, recommended by the national immunization program. This is a multicentric, observational, case-control study. Participants Cases with the disease will be compared to Control Participants, that is, without the disease, regarding the vaccination history for Covid-19.Complementarily, an evaluation of cellular and humoral immunity will be carried out in a sample of both case and control participants, taking into account the vaccination history.

DETAILED DESCRIPTION:
The Covid-19 vaccines currently distributed by the National Immunization Program (NIP) have undergone a rigorous safety and efficacy assessment by the National Surveillance Agency Sanitary prior to the authorization of use in the country. The main objective of vaccination against Covid19 is to reduce its morbidity and mortality and, in the future, to promote the control of transmission from the prevention of symptomatic cases in the general population.

To achieve this goal, however, it is important that the vaccines are administered correctly (according to the vaccination schedule correct application techniques and appropriate storage conditions, for example), in the selected population groups (according to prioritization criteria), with vaccination coverage and selected population groups (according to prioritization criteria), with vaccination coverage and vaccination speeds sufficient for effective control of the disease.That is, there are factors that extrapolate the issues of quality, efficacy and safety evaluated in the pre-registration stages, which are extremely important for the success of immunization programs. Thus, the monitoring of these parameters after large-scale use is essential to ratify the favorable risk-benefit assessment made at the time of decision on the introduction of these vaccines in the NIP.

Regarding the role of vaccines in the prevention and control of target diseases, in addition to data from efficacy and immunogenicity obtained in the controlled situations of clinical trials, it is necessary to extend this assessment to routine situations, i.e., "real life", based on the so-called effectiveness studies. Factors such as storage and administration conditions of these products, issues related to vaccinated populations and individuals may affect the response to vaccines.

Therefore, the monitoring of effectiveness must be continuous, seeking to prove the impact of the vaccines in reducing the occurrence of the disease, as well as generating vaccine immunogenicity data, which can be used in the future as protective inferences in complementary analyses.

Thus, the present research project is a study of the effectiveness of the vaccination whereas the efficacy of licensed vaccines, demonstrated in controlled studies, that needs to be verified in the routine of immunization services throughout the country, with its diversity including different vaccination coverage and circulation of SARS-CoV-2 variants, as well as individual factors, such as age group and presence of comorbidities.

The performance of immunization in susceptible population generates groups exposed and not exposed to the COVID-19 vaccine.

Underlying hypothetical cohorts of vaccinated and unvaccinated cannot be clearly enumerated, and the strategy is to reconstruct the experience of exposure (vaccination) and disease (COVID-19) in this population.

In addition to efficacy data obtained from pre-licensing/authorisation clinical trials and the monitoring of vaccine effectiveness, the main objective of this study, to obtain data on the development of immune response to symptomatic SARS-CoV-2 infection (COVID-19) is of great importance for future immunization actions, especially, the development of future vaccines. In the near future, with the increasing availability of vaccines COVID-19, it will become increasingly difficult (for ethical and programmatic reasons) to conduct trials placebo-controlled clinical trials, which may be replaced by immunogenicity studies.

However, for this, it will be necessary to improve knowledge in relation to the post-infection immune response and also that triggered by vaccination, moving towards the definition of the so-called correlates of serum protection.

In this context, we included in the present case-control study proposal, the establishment of a cohort of cases and controls, grouped according to vaccination history for COVID-19, for follow-up and evaluation of your humoral and cellular immune response.

We understand be an opportunity, based on the identification of virologically confirmed cases and a control with SARS-CoV-2 infection known to be ruled out, observe and describe the humoral and cellular immune response components in these research participants, including duration immunity for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in the study after reading, understanding and signing the informed consent.
* Availability and possibility of being followed up during the follow-up period defined in the study, through visits to research centers, home visits, telephone contacts or other means of digital communication.
* Completing the case or control definitions described below.

Exclusion Criteria:

* Behavioral, cognitive or psychiatric illness that, in the opinion of the responsible investigator or his/her medical representative, affects the participant's ability to understand and comply with the requirements of the study protocol;
* Any other condition that, in the opinion of the responsible investigator or his/her medical representative, may jeopardize the safety or rights of a potential participant or prevent him/her from complying with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants virologically confirmed incident cases of COVID-19 and Control Participants without COVID-19 (no suspected symptomatology and RT-PCR negative for SARS-CoV in two consecutive naso/oropharyngeal swab samples).
Sampling Method: Non-Probability Sample
Enrollment: 3920 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of the vaccination against COVID-19. | 12 months
  Confirmed disease (RT-PCR positive for SARS-CoV-2), according to:the clinical spectrum (of mild disease , moderate to severe) and outcome (disease-related death);according to the vaccine used, the number of doses and the interval rom the last dose to the onset of symptom;according to the presence of comorbidities and medication use; according to Region/State;according to vaccination coverage;according to circulating viral variants.

SECONDARY OUTCOMES:
Assess the humoral and cellular immune response | 15 months
  in vaccinated or unvaccinated cases compared to vaccinated or unvaccinated controls.
Analyze individual factors | 15 months
  including those related to the adaptive immune response (HLA molecules) and genetic aspects, in severe cases/deaths associated with vaccine failures.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Technology in Immunobiology Bio-Manguinhos/Fiocruz, Rio de Janeiro, Brazil